CLINICAL TRIAL: NCT04794335
Title: Pharmacology of Visceral Afferents
Brief Title: Visceral Afferents
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Gold, Professor, University of Pittsburgh
Other Study IDs: STUDY20070343; R01DK107966 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-03-12 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: pain; nociceptor; sensitization
MeSH Terms: conditions — Inflammatory Bowel Diseases; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The only tissue recovered as part of this study is the intestine removed as part of a surgical procedure. Pieces of tissue to be analyzed for protein or mRNA will be stored at -80oC in a laboratory freezer. Tissue will be processed in batches. Any tissue not processed by the end of the 5 year study will be disposed of as medical waste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing resection of intestine for therapeutic purposes: Tissue will be accepted from all eligible donors who consent to having their intestine removed for therapeutic purposes. This tissue would normally be disposed of as medical waste, used for research purposes. The tissue will be studied in the lab in a series of experiments involving GABA agonists and antagonists. Each GABA agonist and/or agonists/antagonist combination will be studied on intestine tissue randomly assigned to one of four groups defined by patient sex (m/f) and the application of inflammatory mediators (+/-). Thus, four groups are needed per GABA agonist and agonist/antagonist combination and seven agonist/antagonist combinations will be tested for a total of 28 experimental groups. But all of these groups will be generated from all patients recruited for the study.

SUMMARY:
The vast majority of what is known about the extrinsic innervation of the visceral was obtained through the study of preclinical models, primarily rats and mice. Given a growing list of important species differences, the investigators wish to determine the extent to which what scientists think they know about the control of visceral afferent excitability learned through the study of rodents holds true for humans. The investigators wish to establish an ex-vivo preparation using intestine surgically removed for the treatment of cancer, ischemia, etc, that would normally be disposed of as medical waste, to study the properties of the extrinsic innervation of the intestine. Tissue will be recovered in the OR, taken back to the lab, and evoked activity in the neurons innervating the intestine will be studied with extracellular recording techniques. Pharmacological approaches will be used to characterize the ion channels/receptors controlling the excitability of visceral afferents. After recording, tissue may be further analyzed with biochemical approaches such as western blot, PCR, and/or flow cytometry.

DETAILED DESCRIPTION:
Visceral pain disorders such as irritable bowel syndrome (IBS) and inflammatory bowel diseases (IBD; Crohn's disease, ulcerative colitis) remain a significant health problem both because of the large number of people who suffer from these disorders and because there are few, if any consistently effective therapeutic interventions. Thus, the goal of this project is to identify novel therapeutic approaches for the treatment of visceral pain.

The sensation of visceral pain is transmitted from visceral structures to the central nervous system via sensory neurons where the increase in pain associated with IBS and IBD is due, at least in part to increases in the excitability of these sensory neurons. Virtually all that scientists know about visceral sensory neurons was learned through the study of non-human species, in particular, rats and mice. A growing body of evidence suggests that many of the discoveries made in these species have failed to translate into more effective treatments because of species differences. To address this gap in knowledge, the investigators have proposed to study human tissue. Based on the investigator's preclinical data, they will start with a focus on GABA receptors, but will also explore other ionotropic receptors (for serotonin and ATP), as well as voltage gated ion channels. The investigators hypothesize that the dearth of effective treatments for visceral pain is due, at least in part, to species differences in the channels controlling the excitability of visceral sensory neurons. Electrophysiological techniques combined with pharmacological approaches will be used for a functional analysis of visceral afferents, and these endpoints will be complimented by biochemical, anatomical, and molecular biological analyses. Electrophysiological analysis of tissue will be performed on the day of surgery. Tissue will be processed and stored for biochemical, anatomical, and molecular biological analyses on the day of surgery, but analyzed once per month if it is possible to recover tissue from two patients per week.

ELIGIBILITY:
Inclusion Criteria:

* This study's inclusion criteria are fairly straightforward: an adult (>18), younger than 85
* Scheduled for abdominal surgery involving the removal of GI tissue for therapeutic purposes
* Meets ASA 1-3 criteria.

Exclusion Criteria:

* Subject <18 years of age.
* Subject declines participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects (>18), younger than 85, scheduled for abdominal surgery involving the removal of GI tissue for therapeutic purposes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Single unit activity in afferents innervating intestine specimen | The presence of activity will be assessed immediately in each specimen recovered, day 1 of surgery.
  The success of this ex vivo study will depend on the ability to record from afferent providing extrinsic innervation to the intestine.
The ability to identify receptive fields of visceral afferents in the intestine | The presence of receptive fields will be assessed immediately in each specimen recovered, day 1 of surgery.
  An electrical search strategy will be used to identify receptive fields in the ex vivo preparation
Pharmacological characterization of isolated visceral afferent | Pharmacological analysis will be performed immediately on each specimen recovered day 1 of surgery.
  The impact of GABAA agonists and/or agonist/antagonist combinations will be assessed in the ex vivo preparation
Changes in threshold of action potential generation in response to inflammatory mediators and/or GABAA agonists or agonist/antagonist combinations. | Excitability will be analyzed immediately on each specimen recovered, day 1 of surgery.
  The pharmacological characterization of isolated units will involve the assessment of changes in activity evoked with stretch of the intestine.

SECONDARY OUTCOMES:
Biochemical characterization of GABAA receptor signaling molecules in human intestine | Tissue for biochemical analysis will be flash frozen on day 1 of surgery.
  Biochemical approaches such as western blot will be used to assess the presence and density of GABAA receptor signaling machinery (receptors, GABA transporters, etc), in human intestine. This analysis will be performed in tissue not used for pharmacological analysis.
Anatomical characterization of GABAA receptor signaling molecules in human intestine | Tissue for anatomical analysis will be immersion fixed on day 1 of surgery.
  Anatomical approaches such as immunohistochemistry will be used to assess the presence and density of GABAA receptor signaling machinery (receptors, GABA transporters, etc), in human intestine. This analysis will be performed in tissue not used for pharmacological analysis.
Molecular biological characterization of GABAA receptor signaling molecules in human intestine | Tissue for molecular biological analysis will be flash frozen on day 1 of surgery.
  Molecular biological approaches such as semi-quantitative PCR will be used to assess the presence and density of GABAA receptor signaling machinery (receptors, GABA transporters, etc), in human intestine. This analysis will be performed in tissue not used for pharmacological analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Gold, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center (UPMC) Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
All data generated from this study will be made publicly available through publications.